CLINICAL TRIAL: NCT01696305
Title: Prospective, Randomized, Double Blind, Multicenter Study for Hyalobarrier ® to Evaluate Anti-adhesive Effect and Safety Compared to Guardix-SG® After Thyroidectomy
Brief Title: Study for Hyalobarrier to Evaluate Anti-adhesive Effect and Safety Compared to Guardix-SG After Thyroidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hyalobarrier_P3
Record Dates: First submitted 2012-09-26; First posted 2012-10-01 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Thyroid Disease
Keywords: Thyroid disease; Hyalobarrier; Thyroidectomy; anti-adhesive effect
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyalobarrier (Experimental): ACP200 (Auto-crosslinked polysaccharide:inner ester of hyaluronic acid) 30mg/ml*10ml/syringe and 5cm-cannula
  Interventions: Device: Hyalobarrier
- Guardix-SG (Active Comparator): Poloxamer/sodium alginate mixture 6g/syringe
  Interventions: Device: Guardix-SG

INTERVENTIONS:
Device: Hyalobarrier
  Arms: Hyalobarrier
Device: Guardix-SG
  Arms: Guardix-SG

SUMMARY:
This study is a randomized, double-blind, active controlled phase 3 trial in the patients with thyroid disease, who will undergo total thyroidectomy (excluding the patients with the patient with the past history of thyroid surgery).

An eligible patient will be randomized and allocated to either the test group (Hyalobarrier) or active-comparator group (Guardix-SG). He/she will undergo marshmallow esophagography in detecting esophageal dysmotility at 6 weeks after study intervention and will be followed for 12weeks.

During the study, both the patients and the observer for the primary and secondary efficacy evaluation will be masked.

Non-inferiority of the test device (Hyalobarrier) compared to the reference device (Guardix-SG) will be confirmed using the primary efficacy outcome,the percentage of normal esophageal transit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female between 18 and 79 years of age
* Patients diagnosed with thyroid disease who will undergo total thyroidectomy
* Naive patients to thyroid surgery
* Given written informed consent
* Childbearing potential female patients who give the consent for contraception during the study

Exclusion Criteria:

* Pregnant or breast-feeding female patients
* Abnormal coagulation panel test
* Clinically abnormal laboratory values
* Inappropriate general health conditions
* Past or current medication history for hyperthyroidism
* Medication with aspirin (or anti-platelet) before surgery
* Current medication with anticoagulants
* Inoperable (thyroidectomy) concurrent diseases
* Concurrent diseases/conditions which will be unable to evaluate the primary and secondary outcomes
* Participating in other interventional clinical trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2012-12; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
The percentage of normal esophageal transit in marshmallow esophagography | 6 Weeks after intervention

SECONDARY OUTCOMES:
Adhesion severity using VAS | Baseline and 1, 6 and 12 weeks
Swallow impairment | Baseline and 1, 6 and 12 weeks
Voice impairment | Baseline and 1, 6 and 12 weeks
voice behavior using Voice Range Profile (VRP) assessment | Baseline and 1, 6 and 12 weeks
Injury of recurrent laryngeal nerve | Baseline and 1, 6 and 12 weeks
Postoperative Sore Throat within 24hours after thyroidectomy | Pre- and Post (0, 24h)-opreation
Adverse Events | during 12 weeks after investigational device use

CONTACTS AND LOCATIONS:
Overall Officials: Hoon Yub Kim, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital; Jae-Bok Lee, M.D., Ph.D., Principal Investigator — Korea University Guro Hospital; Kyoung Sik Park, M.D., Ph.D., Principal Investigator — Konkuk University Medical Center
Locations (3):
- South Korea (3):
  - Konkuk University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul